CLINICAL TRIAL: NCT05234333
Title: COVID-19 Vaccines Induced Malaise: A Retrospective Study and Analysis of the WHO Pharmacovigilance Database
Brief Title: COVID-19 Vaccines Associated Malaise
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20220203
Record Dates: First submitted 2022-02-09; First posted 2022-02-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Vaccine Adverse Reaction
MeSH Terms: interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients presenting a malaise after the vaccination by any vaccine
  Interventions: Drug: SARS-CoV-2 vaccine
- Patients presenting any other adverse event after the vaccination by any vaccine
  Interventions: Drug: SARS-CoV-2 vaccine

INTERVENTIONS:
Drug: SARS-CoV-2 vaccine — SARS-CoV-2 vaccination

SUMMARY:
COVID-19 vaccines induced malaise have recently been reported in the literature. Our study aims to identify risk factors associated with the onset of COVID-19 vaccines induced malaise and to assess if certain COVID-19 vaccines could be more prone to cause malaise compared to influenza vaccines.

To do so we performed a disproportionality analysis adjusted on age class, sex, region and type of reporter in VigiBase®, the WHO pharmacovigilance database, restricted to data from 01/01/2021 to 26/01/2022 to assess the association between all COVID-19 vaccines on the market and malaise. Demographic data were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* all adverse events reported in the WHO pharmacovigilance database

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients
Sampling Method: Non-Probability Sample
Enrollment: 1534706 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
disproportionality analysis in VigiBase® : search for an over-reporting of malaise with COVID-19 vaccines compared to influenza vaccines | from the 01/01/2021 to the 26/01/2022
  case/no case study

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France